CLINICAL TRIAL: NCT02577627
Title: Multi-Centre, Multi-Indication, Two-Stage, Oncological Study to Retrospectively Assess and Prospectively Validate the Predictive Accuracy of PrediCare - a Standalone, Treatment Decision Support Software Device for Predicting Time-to-Progression in Individual Patients Under Standard of Care Treatments
Brief Title: Multi-Indication, Retrospective Oncological Study to Validate the Accuracy in Predicting TTP by PrediCare in Patients Under SOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Optimata Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OPTI-006
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2016-09

CONDITIONS: Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Prostate Cancer; Breast Cancer; Colon Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Prostatic Neoplasms; Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Training Set: The Training Set will be used to calibrate the Predicare models and algorithms and assess its predictive potential in a retrospective manner. Patients data will be collected according to the oncological indications (NSCLC, SCLC, Prostate cancer, Breast cancer and Colon cancer) and the applied treatment protocols, and their data will be integrated and processed by the PrediCare algorithm.
  Interventions: Device: PrediCare
- Validation Set: The Validation Set will be used to validate the prediction power of the device in a prospective manner. The files of patients assigned to Validation Set of the study will be used for the blind prediction of TTP under each specific treatment, based on the baseline individual information. This will be done by inputting into PrediCare the information of each individual patient, available prior to treatment onset (baseline; clinical data, imaging data, histology/cytology, oncomarkers, genetic screening, hematology, biochemistry) for creating a personalized mathematical models and predicting TTP of this specific patient. These predictions will be then compared to the clinically observed TTP for all the patients.
  Interventions: Device: PrediCare

INTERVENTIONS:
Device: PrediCare

SUMMARY:
This is a retrospective observational, open label study to evaluate and prospectively validate in a blind manner the accuracy of predicting treatment outcomes by PrediCare in individual patients with Non-Small Cell Lung Cancer, Small Cell Lung Cancer, Castration-Resistant Prostate Cancer, Breast Cancer & Colon Cancer under the treatment with the mono- and combination drug protocols for the 1st and 2nd line treatment, approved to the market as a Standard of Care

DETAILED DESCRIPTION:
The goals of this study are assessing and validating the accuracy of the PrediCare predictions by comparing them to the actual patients outcome. Study population will be composed of patients diagnosed with advanced stage disease, and divided according to the indications and treatment protocols. Retrospective data collected from patients' files will enable Optimata to compare the PrediCare Technology predictions of the pattern of metastatic and primary tumor growth and dynamics of oncological markers over time with the actual outcomes in each individual patient.

ELIGIBILITY:
Inclusion Criteria:

Lung Cancer (NSCLC):

1. Gender: Female, Male.
2. Age: Eighteen years and older at the start of treatment.
3. Stage: Pathologically or cytologically determined advanced or locally advanced NSCLC at Stage III/IV, adenocarcinoma, OR Pathologically or cytologically determined advanced or locally advanced NSCLC at Stage III/IV, NOS.
4. Lung cancer with measurable disease at the start of treatment.
5. No prior chemotherapy unless used in adjuvant therapy, completed more than 12 month before.
6. Patient has at least one quantitative measurements of at least one lesion in lung (primary tumor or metastasis) before treatment.
7. Patient has at least one quantitative measurements of at least one lesion in lung (primary tumor or metastasis) during or after the treatment.
8. Patient has at least one recorded visit to the treating oncologist before treatment.
9. Patient has at least one recorded visit to the treating oncologist during or after the treatment.
10. Treatment as per SOC for NSCLC.

Lung Cancer (SCLC):

1. Genders Eligible for Study: Female/Male patient.
2. Ages between 18 and older at the start of treatment.
3. Pathologically or cytologically determined advanced or locally advanced SCLC at Stage III/IV.
4. Lung cancer with measurable disease at the start of treatment.
5. No prior chemotherapy unless used in adjuvant therapy, completed more than 12 month ago.
6. Patient has at least one quantitative measurements of at least one lesion in lung (primary tumor or metastasis) before treatment.
7. Patient has at least one quantitative measurements of at least one lesion (primary tumor or metastasis) during or after the treatment.
8. Patient has at least one recorded visit to the treating oncologist before treatment.
9. Patient has at least one recorded visit to the treating oncologist during or after the treatment.
10. Treatment as per SOC for SCLC.

Colon Cancer:

1. Genders Eligible for Study: Female/Male patient.
2. Ages between 18 and older at the start of treatment.
3. Pathologically or cytologically determined advanced or locally advanced Colon Cancer at Stage III/IV
4. Colon cancer with measurable disease at the start of treatment
5. No prior chemotherapy unless used in adjuvant therapy, completed more than 12 month ago,
6. Patient has at least one quantitative measurements of at least one lesion (primary tumor or metastasis) before treatment
7. Patient has at least one quantitative measurements of at least one lesion (primary tumor or metastasis) during or after the treatment.
8. Patient has at least one recorded visit to the treating oncologist before treatment
9. Patient has at least one recorded visit to the treating oncologist during or after the treatment.
10. Treatment as per SOC for Colon cancer

Breast Cancer:

1. Genders Eligible for Study: Female patient.
2. Ages between 18 and older at the start of treatment.
3. Patients must have histologically confirmed breast malignancy that is either:

   * Stage III breast cancer, including inflammatory breast cancer, or
   * Stage IV breast cancer in a complete remission (bone only not allowed unless the bone scan is normal).
4. Breast cancer with measurable disease at the start of treatment.
5. No prior chemotherapy unless used in adjuvant therapy, completed more than 12 month ago.
6. Patient has at least one quantitative measurements of at least one lesion (primary tumor or metastasis) before treatment.
7. Patient has at least one quantitative measurements of at least one lesion (primary tumor or metastasis) during or after treatment.
8. Patient has at least one recorded visit to the treating oncologist before treatment.
9. Patient has at least one recorded visit to the treating oncologist during or after the treatment.
10. Treatment as per SOC for Breast cancer.

Prostate Cancer:

1. Genders Eligible for Study: Male patient.
2. Ages between 18 and older at the start of treatment.
3. Histologically confirmed prostate cancer with progressive metastatic disease based on any of the following:

   1. Rise in PSA - a minimum of 3 consecutive rising levels, with an interval of ≥1 week between each determination. The last determination must have a minimal value of ≥ 2 ng/mL and be determined within two weeks prior to enrolment.
   2. Measurable Disease by transaxial imaging - patients showing new or progressive soft tissue masses on CT or MRI scans as defined by the PCWG2.
   3. Radionuclide bone scan - at least two new metastatic lesions by CT, MRI or by any SOC.
4. Ongoing androgen depletion therapy with a Gonadotropin Releasing Hormone (GnRH) analogue or inhibitor, or orchiectomy (i.e., surgical or medical castration).
5. Patients must have castrate levels of testosterone (<50 ng/dl [1.74 nmol/l]).
6. Patient has at least one recorded visit to the treating oncologist before treatment.
7. Patient has at least one recorded visit to the treating oncologist during or after the treatment.
8. Treatment as per SOC for Prostate cancer.

Exclusion Criteria:

Lung Cancer (NSCLC):

1. History of another malignancy within the previous 2 years except for the following:

1. Adequately treated basal cell or squamous cell skin cancer,
2. Adequately treated Stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 2 years.

Lung Cancer (SCLC):

1. History of another malignancy within the previous 2 years except for the following: Adequately treated basal cell or squamous cell skin cancer,
2. Adequately treated Stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 2 years.

Colon Cancer:

1. History of another malignancy within the previous 2 years except for the following:

1. Adequately treated basal cell or squamous cell skin cancer,
2. Adequately treated Stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 2 years.

Breast Cancer:

1. Patients who have had chemotherapy or radiotherapy within 6 weeks prior to entering the study.
2. History of another malignancy within the previous 2 years except for the following:

   1. Adequately treated basal cell or squamous cell skin cancer,
   2. Adequately treated Stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 2 years.

Prostate Cancer:

1. History of, or current known metastases in the brain or untreated spinal cord compression;
2. History of another malignancy within the previous 2 years except for the following:

   1. Adequately treated basal cell or squamous cell skin cancer,
   2. Adequately treated Stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 2 years.
3. Patients have received prior cytotoxic chemotherapy for Prostate cancer.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from up to about 1000 NSCLC patients' files will be collected. Data from up to about 1000 SCLC patients' files will be collected. Data from up to about 1000 Colon cancer patients' files will be collected. Data from up to about 1000 Breast cancer patients' files will be collected. Data from up to about 1000 Prostate cancer patients' files will be collected.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-01 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint in this study is Time To Progression of disease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marina Kleiman, PhD, Study Director — Optimata Ltd.; Irina Lazarov, MD, Principal Investigator — Soroka University Medical Center; Maya Gottfried, MD, Principal Investigator — Meir Medical Center, Kfar Saba, Israel; Noa Efrat (Ben-Baruch), MD, Principal Investigator — Kaplan Medical Center, Rehovot, Israel; Mor Moskovitz, MD, Principal Investigator — Rambam Medical Center, Haifa, Israel; Avishay Sela, MD, Principal Investigator — Assaf Harofeh Medical Center, Zrifin, Israel; Ronen Brenner, MD, Principal Investigator — Wolfson Medical Center; Hovav Nehushtan, MD, Principal Investigator — Hadassah Medical Center, Jerusalem
Locations (1):
- Optimata Ltd., Bne ‘Atarot, Israel